CLINICAL TRIAL: NCT01239433
Title: Pathophysiologic Changes in the Respiratory System During Therapeutic Interventions
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Espen Rostrup Nakstad, MD, Oslo University Hospital
Other Study IDs: REK S-O, Ref 2010/1340, part B
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- mechanically ventilated patients: ICU patients on mechanical ventilation. Daily endotracheal suctioning performed to reduce secretions. Data recorded during these therapeutic interventions.

SUMMARY:
Airway pressures change during fiberoptic bronchoscopy and endotracheal suctioning. In this study pressure changes are examined in a mechanical lung model and in a population of ICU patients on mechanical ventilation.

DETAILED DESCRIPTION:
Airway pressures change during fiberoptic bronchoscopy and endotracheal suctioning. In this study such pressure changes are examined in a mechanical lung model and in a population of ICU patients on mechanical ventilation. A systematic recording of airway pressures, tidal volumes and blood gases are carried out during ordinary therapeutic procedures requested by the staff physician. No additional study interventions are carried out.

The aim of the project is to examine negative effects of pressure/volume changes.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* on mechanical ventilation
* daily endotracheal suctioning performed

Exclusion Criteria:

* < 18 years of age
* non-invasive ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the Intensive Care Unit (ICU) on mechanical ventilation where daily endotracheal suctioning is performed to remove secretions.
  Most of the patients have ARDS/ ALI.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Intrabronchial airway pressure | 2013

CONTACTS AND LOCATIONS:
Overall Officials: Espen R Nakstad, MD, Principal Investigator — Oslo University Hospital - Ulleval, Norway; Helge Opdahl, MD, PhD, Study Director — Ullevaal University Hospital
Locations (1):
- Oslo University Hospital - Ulleval, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Undecided